CLINICAL TRIAL: NCT04004065
Title: A Phase 2, Two-Part, Multiple-Ascending-Dose Study of SRP-5051 for Dose Determination, Then Dose Expansion, in Patients With Duchenne Muscular Dystrophy Amenable to Exon 51-Skipping Treatment
Brief Title: Two-Part Study for Dose Determination of Vesleteplirsen (SRP-5051) (Part A), Then Dose Expansion (Part B) in Participants With Duchenne Muscular Dystrophy Amenable to Exon 51-Skipping Treatment
Acronym: MOMENTUM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated following review of safety data.
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5051-201; 2019-000601-77 (EudraCT Number)
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; Duchenne; Dystrophy; Dystrophin; Exon Skipping; Ambulatory; Duchenne Muscular Dystrophy; Exon 51; Nonambulatory; Pediatric; Peptide-conjugated phosphorodiamidate morpholino oligomer (PPMO)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Vesleteplirsen (Experimental): Participants received escalating dose levels of vesleteplirsen, every 4 weeks, via intravenous (IV) infusion for up to 75 weeks during Part A. Once the doses have been selected for Part B, all participants who have completed Part A will transition to Part B.
  Interventions: Drug: Vesleteplirsen
- Part B: Vesleteplirsen (Experimental): Participants received vesleteplirsen at the doses selected based on data from Part A every 4 weeks, via IV infusion, for up to 5 years. This included the participants who rolled over from Part A, as well as the additional participants who enrolled at the beginning of Part B.
  Interventions: Drug: Vesleteplirsen

INTERVENTIONS:
Drug: Vesleteplirsen — Vesleteplirsen injection, for IV use
  Other Names: SRP-5051

SUMMARY:
This study will be comprised of 2 parts: 1) Part A (Multiple Ascending Dose [MAD]) will be conducted to evaluate the safety and tolerability of vesleteplirsen at MAD levels to determine the maximum tolerated dose (MTD), and 2) Part B will be conducted to further evaluate the vesleteplirsen doses selected in Part A. Participants enrolling in Part B will be those who completed Part A or Study 5051-102 (NCT03675126) and meet applicable eligibility criteria for Part B, as well as additional participants who meet applicable eligibility criteria for enrollment at the beginning of Part B.

ELIGIBILITY:
Inclusion Criteria for participants previously treated with Vesleteplirsen:

- Has received prior Vesleteplirsen treatment in Part A of this study or in Study 5051-102.

Exclusion Criteria for participants previously treated with Vesleteplirsen and new participants enrolling into Part B:

- Presence of other clinically significant illness, including cardiac, pulmonary, hepatic, renal, hematologic, immunologic, or behavioral disease, or infection or malignancy or any other condition that, in the Investigator's opinion, could interfere with participation in the trial.

Inclusion Criteria for treatment-naïve participants enrolling into Part B:

* Has a genetic diagnosis of Duchenne muscular dystrophy (DMD) and an out-of-frame deletion mutation of the DMD gene amenable to exon 51-skipping treatment.
* Has been on a stable dose of oral corticosteroids for at least 12 weeks prior to study drug administration and the dose is expected to remain constant throughout the study (except for modifications to accommodate changes in weight), or has not received corticosteroids for at least 12 weeks prior to study drug administration.
* Has stable pulmonary function (forced vital capacity [FVC] ≥40% of predicted and no requirement for nocturnal ventilation).

Exclusion Criteria for treatment-naive participants enrolling into Part B:

* History of hypomagnesemia within 12 weeks prior to Screening.
* Initiation or change of dosing (except for modifications to accommodate changes in weight or changes in standard of care) within 12 weeks prior to Screening for any of the following: angiotensin-converting enzyme inhibitors, angiotensin receptor-blocking agents, β-blockers, or potassium.
* Initiation or change of dosing within 12 weeks prior to Screening for over-the-counter preparations, such as herbal/nonherbal supplements, vitamins, minerals, and homeopathic preparations.
* Has a left ventricular ejection fraction (LVEF) <40.0% based on an echocardiogram (ECHO) performed within 12 weeks prior to Screening or at the Screening Visit.
* Treatment with any exon 51-skipping therapy within 4 weeks prior to Screening, or with any experimental gene therapy for the treatment of DMD at any time.

Other inclusion/exclusion criteria apply.

Ages: 7 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Part A: Incidence of Adverse Events (AEs) | Part A: Baseline up to 75 weeks
Part B: Change From Baseline in Dystrophin Protein Level at Week 28 | Part B: Baseline, Week 28

SECONDARY OUTCOMES:
Part A: Pharmacokinetics (PK): Plasma Concentration of Vesleteplirsen | Pre-dose and at multiple time points (up to 32 hours) after end of infusion
Part A: PK: Urine Concentration of Vesleteplirsen | Pre-dose and at multiple time periods (up to 48 hours) after end of infusion
Part B: Change From Baseline in Exon-Skipping Levels at Week 28 | Part B: Baseline, Week 28
Part B: Incidence of Adverse Events (AEs) | Part B: Baseline up to Week 304
Part B: PK: Plasma Concentration of Vesleteplirsen | Part B predose and at multiple timepoints (up to 48 hours) after end of infusion
Part B: PK: Urine Concentration of Vesleteplirsen | Part B predose and at multiple timepoints (up to 48 hours) after end of infusion
Part B: Change from Baseline in Percent Dystrophin-Positive Fibers (PDPF) and Mean Intensity, as Measured by Immunofluorescence Assay at Week 28 | Part B: Baseline, Week 28

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (25):
- United States (11):
  - University of California Davis Health, Sacramento, California
  - Connecticut Children's, Farmington, Connecticut
  - Northwest Florida Clinical Research Group, LLC, Gulf Breeze, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center Research Inst., Kansas City, Kansas
  - University of Massachusetts, Worcester, Massachusetts
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Austin Neuromuscular Center, Austin, Texas
  - Children's Health Ambulatory Pavilion, Dallas, Texas
  - Seattle Children's, Seattle, Washington
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Children's Hospital - London Health Sciences Centre (LHSC), London, Ontario, Canada
- Germany (2):
  - University of Essen - Children's Hospital, Essen
  - Klinikum der Universität München, Munich
- Italy (2):
  - Fondazione Policlinico Universitario A Gemelli, Rome
  - A.O.U. Citta della Salute e della Scienza di Torino - SS Malattie Neuromuscolari, Department of Neurosciences, Torino
- Leiden University Medical Center, Leiden, Netherlands
- Spain (2):
  - Hospital Sant Joan de Déu. U.B., Barcelona
  - Hospital Universitari I Politecnic La Fe de Valencia, Valencia
- United Kingdom (4):
  - Alder Hey Children's NHS Foundation Trust, Liverpool, Lancashire
  - Royal Hospital for Children (Glasgow), Glasgow
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Oxford University Hospial NHS Foundation Trust, John Radcliffe Hospital, Oxford